CLINICAL TRIAL: NCT04631146
Title: Efficacy and Safety of Camrelizumab for Chinese NSCLC Patients: a Retrospective, Observational, Multicenter Real-World Study
Brief Title: Efficacy and Safety of Camrelizumab in Real-World Study
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Guangdong Association of Clinical Trials (Other)
Responsible Party: Sponsor
Other Study IDs: CTONG2004
Record Dates: First submitted 2020-10-26; First posted 2020-11-17 (Actual); Last update posted 2020-11-17 (Actual); Status verified 2020-10

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — camrelizumab

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Camrelizumab-treated advanced NSCLC: Patients with advanced non-small cell lung cancer treated with camrelizumab. Dosage form, dosage, frequency and duration of camrelizumab is determined according to the investigator's actual clinical practice.
  Interventions: Drug: Camrelizumab

INTERVENTIONS:
Drug: Camrelizumab — PD-1 inhibitors
  Other Names: SHR-1210

SUMMARY:
This observational real-world study is designed to evaluate the efficacy and safety of camrelizumab for the treatment of Chinese NSCLC patients.

DETAILED DESCRIPTION:
Camrelizumab is a humanized antibody for cancer immunotherapy. The National Medical Products Administration (NMPA, China) approved camrelizumab as a first-line treatment of certain patients with NSCLC.

This is a multicenter non-interventional study, NSCLC patients who have been treated with camrelizumab will be included. The main objective of this study is to evaluate the efficacy and safety of camrelizumab in the clinical practice.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old;
2. Histopathological diagnosed confirmed non-small cell lung cancer;
3. Have received at least one camrelizumab injection between August 1, 2019 and December 31, 2020;
4. Traceable cases.

Exclusion Criteria:

1. Patients who have received other immunotherapy at the same time;
2. Patients who were participating in other intervention studies;
3. Patients with other malignant tumors;
4. The researcher believes that the patient is not suitable to participate in this study with any other conditions .

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Total 450 patients who have received camrelizumab with NSCLC will be enrolled. The patients should be registered consecutively in each site.
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2020-11-30 (Estimated); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
pCR | From August 1, 2019 to June 31, 2021
  Neoadjuvant therapy population: pathological complete response rate (pCR).
R0 resection rate. | From August 1, 2019 to June 31, 2021
  Neoadjuvant therapy population: R0 resection rate.
ORR | From August 1, 2019 to June 31, 2021
  Advanced non-small cell lung cancer: objective response rate (ORR).
6-month PFS% | From August 1, 2019 to June 31, 2021
  Advanced non-small cell lung cancer: 6-month progression-free survival rate (PFS%).

SECONDARY OUTCOMES:
MPR | From August 1, 2019 to June 31, 2021
  Neoadjuvant population: main pathological response rate (MPR)
operative rate | From August 1, 2019 to June 31, 2021
  Neoadjuvant population: operative rate
perioperative mortality | From August 1, 2019 to June 31, 2021
  Neoadjuvant population: perioperative mortality
incidence of major postoperative complications | From August 1, 2019 to June 31, 2021
  Neoadjuvant population: incidence of major postoperative complications (within 30 days after surgery).
iORR | From August 1, 2019 to June 31, 2021
  First-line combined treatment population: median treatment cycle number, intracranial objective response rate (iORR) in patients with brain metastasis.
iPFS | From August 1, 2019 to June 31, 2021
  First-line combined treatment population: median treatment cycle number, intracranial progression-free survival (iPFS) in patients with brain metastasis.
AE | From August 1, 2019 to June 31, 2021
  Safety of the general population: Adverse Events (AE).
SAE | From August 1, 2019 to June 31, 2021
  Safety of the general population: Serious Adverse Events (SAE).

CONTACTS AND LOCATIONS:
Overall Officials: Wu Yilong, Doctor, Principal Investigator — Guangdong Lung Cancer Institute, Guangdong General Hospital, Guangdong Academy of Medical Sciences
Locations (1):
- Guangdong Lung Cancer Institute, Guangdong General Hospital, Guangdong Academy of Medical Sciences, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided